CLINICAL TRIAL: NCT03592355
Title: Virtual Visits at Brigham and Women's Hospital: A Randomized Controlled Trial
Brief Title: Virtual Visits at Brigham and Women's Hospital
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19 pandemic
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Levine, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018P000452
Record Dates: First submitted 2018-05-14; First posted 2018-07-19 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure; Hypertension; Diabetes Mellitus; Stroke; BPH; Hyperlipidemia
Keywords: virtual care; virtual visit; telemedicine
MeSH Terms: conditions — Heart Failure; Hypertension; Diabetes Mellitus; Stroke; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Clinicians slated for virtual visit rollout will be randomized (stratified by department) to either receive immediate virtual visit on-boarding (intervention arm) or delayed (3-months later) virtual visit on-boarding (control arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): If enrolled in the intervention arm, the following steps will occur:
  * The Brigham Health Virtual Care team will work with the clinician toward immediate on-boarding (software training, hardware setup, technical support) as per their usual process.
  * The clinician will schedule virtual visits as s/he and/or her/his department see fit. Virtual visits occur on an already-in-use Partners- and Brigham-approved video platform.
  Interventions: Other: Virtual Visit
- Control (No Intervention): If enrolled in the control arm, the following steps will occur:
  * Three months from the time of the follow-up email, the Brigham Health Virtual Care team will work with the clinician toward immediate on-boarding (software training, hardware setup, technical support) as per their usual process.
  * The clinician will schedule virtual visits as s/he and/or her/his department see fit. Virtual visits occur on an already-in-use Partners- and Brigham-approved video platform.

INTERVENTIONS:
Other: Virtual Visit — Clinicians will have a synchronous video visit with their patients.
  Arms: Intervention

SUMMARY:
Clinicians slated for virtual visit rollout will be randomized (stratified by department) to either receive immediate virtual visit on-boarding (intervention arm) or delayed (3-months later) virtual visit on-boarding (control arm). The investigators plan to enroll no more than 200 clinicians.

Any clinician in a department selected by the Brigham Health Virtual Care team for access to virtual visits is eligible, unless s/he saw less than 20 patients monthly over the last 6 months.

The Brigham Health Virtual Care team will onboard all clinicians and provide virtual visit support as per their usual protocol. The primary study endpoint is third-available appointment, a well-adopted measure of access. Other secondary endpoints revolve around continuity, efficiency, utilization, safety, cost, and patient experience.

DETAILED DESCRIPTION:
If enrolled in the intervention arm, the following steps will occur:

* The clinician will receive the intervention arm follow-up email ("Follow-up Email - Intervention" in the Appendix).
* The Brigham Health Virtual Care team will work with the clinician toward immediate on-boarding (software training, hardware setup, technical support) as per their usual process.
* The clinician will schedule virtual visits as s/he and/or her/his department see fit. Virtual visits occur on an already-in-use Partners- and Brigham-approved video platform (attached).

If enrolled in the control arm, the following steps will occur:

* The clinician will receive the control arm follow-up email ("Follow-up Email - Control" in the Appendix).
* Three months from the time of the follow-up email, the Brigham Health Virtual Care team will work with the clinician toward immediate on-boarding (software training, hardware setup, technical support) as per their usual process.
* The clinician will schedule virtual visits as s/he and/or her/his department see fit. Virtual visits occur on an already-in-use Partners- and Brigham-approved video platform (attached).

The investigators plan to follow patients of both clinician cohorts for a total of 6-months. The investigators will perform retrospective review of patient electronic health records and patients will receive a redcap survey (attached), an evaluation mechanism already employed by the Virtual Care team.

Again, aside from the initial randomization and retrospective data collection and analysis, all of the above would have occurred irrespective of this research protocol.

ELIGIBILITY:
Inclusion Criteria:

* Clinician whose department is chosen for virtual visit rollout

Exclusion Criteria:

* Clinician who saw on average fewer than 20 patients monthly over the past 6 months
* Clinician who opts out of virtual visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Days until third available appointment | Through study completion, an average of 6 months
  Number of days until the third available routine appointment, obtained at 12 o'clock each Friday (embargoed appointments not included). The mean of all of the weeks is a clinician's average number of days until the third available routine appointment.

SECONDARY OUTCOMES:
Days until first available appointment | Through study completion, an average of 6 months
  Number of days until the next available routine appointment, obtained at 12 o'clock each Friday (embargoed appointments not included). The mean of all of the weeks is a clinician's average number of days until the next available routine appointment.
Future capacity: percentage of open appointment slots | Through study completion, an average of 6 months
  Percentage of appointment slots that are open and available for booking patients over the next four weeks, obtained at 12 o'clock each Friday (embargoed appointments not included). The mean of all of the weeks is a clinician's future capacity.
Frequency of visits with the usual provider of care | Through study completion, an average of 6 months
  Ratio of the number of visits to the most frequently seen provider to the total number of visits to all providers obtained each month. The mean of all of the months is a clinician's ratio.
Continuity of care index | Through study completion, an average of 6 months
  The number of visits to each individual physician divided by the total number of visits the patient had overall obtained each month. The mean of all of the months is the continuity of care index
No show rate | Through study completion, an average of 6 months
  Ratio of the number of no-show visits to total visit slots obtained each week. The mean of all of the weeks is a clinician's no show rate.
Visit time | Through study completion, an average of 6 months
  In-person: face time with patient per pertinent EHR fields, obtained each week. The mean of all of the weeks is a clinician's visit time.
  Virtual: enter virtual waiting room to video stops, obtained each week. The mean of all of the weeks is a clinician's visit time.
Clinician volume per hour | Through study completion, an average of 6 months
  Patients seen per hour, calculated at the end of the study.
Clinician volume per day | Through study completion, an average of 6 months
  Patients seen per day, all calculated at the end of the study.
Clinician volume per month | Through study completion, an average of 6 months
  Patients seen per month, all calculated at the end of the study.
Clinician volume per 6 months | Through study completion, an average of 6 months
  Patients seen per 6 months, all calculated at the end of the study.
Slot utilization | Through study completion, an average of 6 months
  Ratio of used slots to total slots, obtained each week. The mean of all of the weeks is a clinician's slot utilization.
Number of primary care visits | Through study completion, an average of 6 months
  Number of primary care visits
Number of specialist visits | Through study completion, an average of 6 months
  Number of specialist visits
Number of emergency department visits | Through study completion, an average of 6 months
  Number of emergency department visits
Number of inpatient admissions | Through study completion, an average of 6 months
  Number of inpatient admissions
Number of imaging studies | Through study completion, an average of 6 months
  Number of imaging studies ordered
Number of labs ordered | Through study completion, an average of 6 months
  Number of laboratory studies ordered
Number of medications prescribed | Through study completion, an average of 6 months
  Number of medications prescribed
Patient Experience | Sent electronically within 1 week of the in-person or virtual visit
  Brigham Health Virtual Care team survey sent to participating patients
Revenue from virtual or in-person visit | Through study completion, an average of 6 months
  Revenue garnered by an individual clinician for her/his clinical activity, calculated per hour and per 6 months (denominator: total clinical hours worked).

CONTACTS AND LOCATIONS:
Overall Officials: David Levine, MD, MPH, MA, Principal Investigator — Principal Investigator
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wootton R. Twenty years of telemedicine in chronic disease management--an evidence synthesis. J Telemed Telecare. 2012 Jun;18(4):211-20. doi: 10.1258/jtt.2012.120219. PMID 22674020
- [Background] McLean S, Sheikh A, Cresswell K, Nurmatov U, Mukherjee M, Hemmi A, Pagliari C. The impact of telehealthcare on the quality and safety of care: a systematic overview. PLoS One. 2013 Aug 19;8(8):e71238. doi: 10.1371/journal.pone.0071238. eCollection 2013. PMID 23977001
- [Background] Dorsey ER, Topol EJ. State of Telehealth. N Engl J Med. 2016 Jul 14;375(2):154-61. doi: 10.1056/NEJMra1601705. No abstract available. PMID 27410924